CLINICAL TRIAL: NCT01070082
Title: Pain Associated With ICU Procedures: An International Study
Brief Title: Europain®: A Study of Procedural Pain
Acronym: Europain®
Status: Completed | Type: Observational
Sponsor: Saint-Louis Hospital, Paris, France (Other)
Collaborators: European Society of Intensive Care Medicine (Other)
Responsible Party: Dr. Kathleen Puntillo, Medical ICU, Saint-Louis Hospital, Paris, France
Other Study IDs: 09-066
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2010-04

CONDITIONS: Pain
Keywords: adult ICU patients; procedural pain; pain intensity; pain distress; pain behaviors; pain; ICU procedures
MeSH Terms: conditions — Pain; Pain, Procedural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adult ICU patients undergoing procedure

SUMMARY:
Pain associated with procedures performed on adult ICU patients is ubiquitous and the subject of research attention.While there is growing evidence about the prevalence, characteristics and measurement of procedural pain in ICUs, most of this evidence has been derived from English-speaking patients in the United States who were able to verbally report the intensity and distress of this pain. Frequently performed procedures include turning,chest tube removal,wound care/wound dressing change,endotracheal suctioning,central catheter insertion(arterial/venous, have been a focus for research. Other potentially painful procedures, including lumbar puncture and physiotherapy,are numerous and have not been systematically studied in adults.

Patients unable to verbally report their pain have not been able to participate in procedural pain studies, which has limited the generalizability of study results to a narrow population of ICU patients.

The Specific Aims of this proposed European-based, international study of ICU patients undergoing selected procedures are to:

* Describe patient self-reports of pain intensity and distress
* Describe the behaviors exhibited by patients during a procedure, comparing the behaviors exhibited by those able versus unable to self-report pain intensity and pain distress
* Examine predictors of amount of pain intensity, behavioral responses, and analgesic use related to procedures such as gender, age, language spoken, country, and type of hospital.

Validated pain intensity, pain distress, and behavioral observation instruments will be methodically translated into the predominant languages spoken in our international study sites; research and training packets similar to those developed in a large, multisite study in the United States will be developed and provided to data collection sites; and data collection will occur over a 6-month period of time. Study data will be analyzed and disseminated at international meetings and in publications.

DETAILED DESCRIPTION:
Procedures to be studied are the following:

* TURNING (moving side to side in bed)
* POSITIONING (moving up or down in bed)
* MOBILIZATION (getting out of bed or chair)
* RESPIRATORY EXERCISES (cough, deep breathe)
* PERIPHERAL BLOOD DRAW (insertion of catheter into vein in order to draw out blood)
* PERIPHERAL IV INSERTION (insertion of catheter into vein in order to give medications or fluids)
* ARTERIAL LINE INSERTION (insertion of arterial catheter for blood pressure monitoring and arterial blood draws)
* ENDOTRACHEAL SUCTIONING (insertion of suction catheter into endotracheal tube in order to aspirate secretions)
* TRACHEAL SUCTIONING (insertion of suction catheter into a tracheostomy in order to aspirate secretions)
* CHEST TUBE REMOVAL (removal of a tube from the mediastinum or plural space)
* WOUND DRAIN REMOVAL (removal of a drain from a wound such as a drain inserted during abdominal surgery)
* WOUND CARE (i.e., cleaning, dressing change)

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years of age or older
* Patient's primary language is of the country where the evaluation is performed
* Patient meets IRB/Central EC requirements of the institution/ country where the evaluation is performed
* Patient is receiving one of the study's procedures as part of standard care

Exclusion Criteria:

* Patient's condition is very unstable at this time
* Patient is receiving neuromuscular blocking medications
* Patient has a disease or condition, such as Guillain-Barre, that alters sensory transmission proximal to procedure site
* Patient has a disease or condition that would confuse the behavioural assessment, such as decerebrate posturing
* Patient is, or probably is, delirious

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients who are undergoing any of the study procedures and consent to participate. Adults age 18 and over will be eligible for the study if they meet study inclusion criteria and don't meet any exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 5150 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 1 minute
  Pain intensity will be measured through the use of a 0 -10 numeric rating scale (NRS), with higher numbers meaning greater pain intensity.
Pain Distress | 1 minute
  Negative emotional responses to painful stimuli (i.e., distress) can be measured separate from pain intensity. Since pain is defined as an unpleasant sensory and emotional experience, it is expected that patients in this study will be able to report pain distress associated with procedures as well as pain intensity. Pain distress will be measured with a 0-10 NRS, where higher numbers connote a greater degree of distress.
Pain Behaviors | 1 minute
  Observing behavioral indices of pain is another aspect of measuring pain. When patients are undergoing painful procedures, complex neural interactions from the noxious stimulus cause a behavioral response.

CONTACTS AND LOCATIONS:
Overall Officials: kathleen Puntillo, RN DNSc FAAN, Principal Investigator — Medical ICU, Saint-Louis Hospital, Paris, France
Locations (1):
- Medical ICU, Saint-Louis Hospital, Paris, France

REFERENCES:
- [Derived] Puntillo KA, Max A, Timsit JF, Vignoud L, Chanques G, Robleda G, Roche-Campo F, Mancebo J, Divatia JV, Soares M, Ionescu DC, Grintescu IM, Vasiliu IL, Maggiore SM, Rusinova K, Owczuk R, Egerod I, Papathanassoglou ED, Kyranou M, Joynt GM, Burghi G, Freebairn RC, Ho KM, Kaarlola A, Gerritsen RT, Kesecioglu J, Sulaj MM, Norrenberg M, Benoit DD, Seha MS, Hennein A, Periera FJ, Benbenishty JS, Abroug F, Aquilina A, Monte JR, An Y, Azoulay E. Determinants of procedural pain intensity in the intensive care unit. The Europain(R) study. Am J Respir Crit Care Med. 2014 Jan 1;189(1):39-47. doi: 10.1164/rccm.201306-1174OC. PMID 24262016